CLINICAL TRIAL: NCT00040794
Title: ZD1839 (NSC #715055, IND #61187) With Induction Paclitaxel And Carboplatin Followed By Either Radiation Or Concomitant Radiation With Weekly Paclitaxel And Carboplatin In Stage III Non-Small Cell Lung Cancer, A Phase II Study
Brief Title: Combination Chemotherapy, Radiation Therapy, and Gefitinib in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02821; CALGB-30106; CDR0000069407; U10CA031946 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin; Gefitinib; Radiotherapy; Radiation

ARMS (2):
- Stratum I (gefitinib, radiotherapy) (Experimental): Patients receive gefitinib orally (PO) daily for 7 weeks. Patients also undergo concurrent radiotherapy once daily 5 days a week for 7 weeks.
  Patients then receive gefitinib PO daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Radiation: radiation therapy; Other: laboratory biomarker analysis
- Stratum II (gefitinib, radiotherapy, chemotherapy) (Experimental): Patients receive gefitinib and radiotherapy as in stratum I concurrently with paclitaxel IV over 1 hour followed by carboplatin over 30 minutes once weekly for 7 weeks.
  Patients then receive gefitinib PO daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: gefitinib; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Stratum II (gefitinib, radiotherapy, chemotherapy)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Stratum II (gefitinib, radiotherapy, chemotherapy)
Drug: gefitinib — Given PO
  Other Names: Iressa; ZD 1839
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II clinical trial studies how well combining different regimens of chemotherapy and gefitinib with radiation therapy work in treating patients with stage III non-small cell lung cancer. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies such as gefitinib may interfere with the growth of tumor cells and slow the growth of non-small cell lung cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving different regimens of combination therapy together with gefitinib and radiation therapy may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether ZD1839 (gefitinib) at 250 mg orally every day administered concomitantly with radiotherapy after induction treatment consisting of paclitaxel, carboplatin, and ZD1839 among patients with inoperable stage III non-small cell lung cancer and Common Terminology Criteria (CTC) performance status 2 or poor risk performance status 0-1 is tolerable.

II. To determine whether ZD1839 at 250 mg orally every day administered concomitantly with paclitaxel, carboplatin, and radiation after induction treatment consisting of paclitaxel, carboplatin, and ZD1839 among patients with inoperable stage III non-small cell lung cancer and CTC performance status 0-1 is tolerable.

III. To determine the overall response rate, failure-free survival, and survival after treatment with induction chemotherapy with daily ZD1839, concomitant radiotherapy and daily ZD1839, and post-radiotherapy single agent daily ZD1839 among patients with CTC performance status 2 or poor risk performance status 0-1 and inoperable stage III non-small cell lung cancer.

IV. To determine the overall response rate, failure-free survival, and survival after treatment with induction chemotherapy and daily ZD1839, concomitant chemoradiotherapy and daily ZD1839, and post-radiotherapy single agent daily ZD1839 among patients with CTC performance status 0-1 and inoperable stage III non-small cell lung cancer.

V. To determine if elevated circulating epidermal growth factor receptor (EGFR) levels prior to treatment, as determined by either quantitative polymerase chain reaction (PCR) or direct enzyme-linked immunosorbent assay (ELISA) measurement, may predict for response to therapy with EGFR inhibitors.

OUTLINE:

All patients receive induction therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses. Patients then receive therapy based on their assigned stratum.

STRATUM I: Patients receive gefitinib orally (PO) daily for 7 weeks. Patients also undergo concurrent radiotherapy once daily 5 days a week for 7 weeks.

STRATUM II: Patients receive gefitinib and radiotherapy as in stratum I concurrently with paclitaxel IV over 1 hour followed by carboplatin over 30 minutes once weekly for 7 weeks.

Patients then receive gefitinib PO daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-small cell lung cancer (NSCLC), including squamous cell carcinoma, adenocarcinoma (including bronchoalveolar cell), and large cell anaplastic carcinoma (including giant and clear cell carcinomas)
* ELIGIBLE DISEASE STAGES: Inoperable IIIA and selected IIIB

  * Generally, patients entered must be considered unresectable or inoperable; patients with T1 or T2, N2 disease are eligible; patients with T3, N2 or T4, N0-N2 disease are eligible if based on the closeness to the carina, invasion of the mediastinum or invasion of the chest wall; patients with T3, N0-N1 disease are not eligible; patients must be M0 (M1 patients are not eligible)

    * Patients with direct invasion of vertebral body are ineligible
    * Patients with tumors adjacent to a vertebral body are eligible, unless there is demonstrable bone invasion, as long as all gross disease can be encompassed in the radiation boost field in accordance with the homogeneity criteria
    * Patients with contralateral mediastinal disease (N3) are eligible if all gross disease can be encompassed in the radiation boost field in accordance with the homogeneity criteria; patients with scalene, supraclavicular, or contralateral hilar node involvement are ineligible
    * Patients with a pleural effusion, which is a transudate, cytologically negative and non-bloody, are eligible if the radiation oncologist feels the tumor can be encompassed within a reasonable field of radiotherapy. Patients with exudative, bloody, or cytologically malignant effusions are not eligible; if a pleural effusion can be seen on the chest computed tomography (CT) but not on chest x-ray (CXR) and is too small to tap, the patient will be eligible; a pleural effusion appearing only after a thoracotomy or other invasive thoracic procedure was attempted will not make a patient ineligible
* PATIENTS MUST HAVE MEASURABLE DISEASE

  * Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as ≥10 mm with spiral CT scan
  * Lesions that are not considered measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area
* PRIOR THERAPY

  * >= 2 weeks since formal exploratory thoracotomy.
  * No prior chemotherapy or radiation therapy for NSCLC
* CTC performance status 0-2
* No "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Non-pregnant and non-nursing because of significant risk to the fetus/infant
* No patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No patients with chronic gastrointestinal disorders including liver disease, diarrheal or emetic disorders, or malabsorptive conditions which could worsen toxicity or limit efficacy of ZD1839
* No cytochrome P450 3A4 (CYP3A4) inducers within 7 days prior to starting protocol therapy and while on protocol treatment. CYP3A4 inducers: phenytoin, carbamazepine, barbiturates, rifampicin, dexamethasone, and St John's Wort; single doses of dexamethasone used as an antiemetic are permitted
* No human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy
* Granulocytes >= 1,500/ul
* Platelets >= 100,000/ul
* Calculated creatinine clearance >= 20 cc/min
* Bilirubin < 1.5 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2002-05; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Overall survival (Stratum I) | From randomization until death or last known follow-up, assessed up to 10 months
  Kaplan-Meier curves will be used to describe overall survival in each stratum.
Overall survival (Stratum I) | From randomization until death or last known follow-up, assessed up to 13 months
  Kaplan-Meier curves will be used to describe overall survival in each stratum.
Overall survival (Stratum II) | From randomization until death or last known follow-up, assessed up to 14.5 months
  Kaplan-Meier curves will be used to describe overall survival in each stratum.
Toxicity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 3 years
  The frequency of toxicity occurrence will be tabulated by the most severe occurrence.
Failure-free survival | Time between randomization and disease progression, death, or last known follow-up, assessed up to 3 years
  Kaplan-Meier curves will be used to describe failure-free survival in each stratum. Within each treatment group, the pattern of treatment failure (local, distant, regional) will be summarized.
Response to induction treatment | Up to 3 years
  Summarized by treatment group. Exact binomial confidence intervals will be computed for these response rates.
Overall response | Up to 3 years
  Overall response to the full treatment regimen will be summarized by treatment group. Exact binomial confidence intervals will be computed for these response rates.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States